CLINICAL TRIAL: NCT07182006
Title: Movement as Medicine: Can a Single Bout of Aerobic Exercise Elicit Exercise-induced Hypoalgesia in Youth With and Without Chronic Pain Syndromes?
Brief Title: Exercise as Medicine for Pediatric Chronic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Julie Shulman, Physical Therapy Scientist, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P00049713
Record Dates: First submitted 2025-09-09; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Child; Adolescent
Keywords: aerobic exercise; chronic pain; pediatric; quantitative sensory testing; endogenous pain modulation
MeSH Terms: conditions — Chronic Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Youth with chronic pain and healthy controls will complete all study outcomes in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Youth with Chronic Pain Syndromes (Experimental): Youth with chronic pain will undergo quantitative sensory testing before and immediately after a single bout of intense aerobic exercise.
  Interventions: Behavioral: Aerobic Exercise
- Youth without Chronic Pain Syndromes (Active Comparator): Youth without chronic pain will undergo quantitative sensory testing before and immediately after a single bout of intense aerobic exercise. They will serve as a control group to determine if the intervention has different effects between groups.
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Submaximal cardiovascular endurance testing on a treadmill

SUMMARY:
Youth with chronic pain struggle to go to school, play sports, or spend time with friends and family due to pain. Medications are often ineffective, and aerobic exercise may improve both pain sensitivity and participation in valued life activities. This study will be the first to examine the impact of a single session of intense aerobic exercise on pain sensitivity measures in youth with and without chronic pain syndromes to help determine if aerobic exercise can improve pain and functioning.

DETAILED DESCRIPTION:
Pediatric chronic pain syndromes that occur in 11-38% of youth commonly impact participation in school, family, and recreational activities. Pediatric chronic pain and disability can persist into adulthood if left untreated. Central sensitization is an overarching mechanism of pediatric and adult chronic pain syndromes and is conceptualized as an imbalance in the facilitatory and inhibitory pathways that control pain signal traffic in the central nervous system. Aerobic exercise commonly recommended to improve pain and disability, but empirical evidence is lacking. Exercise-induced hypoalgesia (EIH) is a proposed mechanism by which aerobic exercise improves pain sensitivity and is characterized by improved pain sensitivity immediately following exercise. To date, EIH has not been studied in youth with chronic pain syndromes. Insights may reveal potential treatment targets and mechanisms by which aerobic exercise can improve pain and quality of life among youth suffering from chronic pain. This study aims to 1) evaluate and compare EIH responses in youth with and without chronic pain and 2) identify potential biopsychosocial contributors to EIH. The investigators hypothesize that EIH is robust in pain-free youth, and present but attenuated in youth with chronic pain (Aim 1) and that unhelpful beliefs about pain will attenuate the effects of exercise on pain sensitivity (Aim 2). Results from this study will provide highly relevant data to design a clinical trial studying the effects of chronic aerobic exercise on pain and disability in these youth. Identification of effective nonpharmacologic treatments for chronic pain, such as exercise, may also reduce dependence on prescription medications and improve child health.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary chronic pain syndrome

Exclusion Criteria:

* Allodynia (pain with light touch) at testing sites (non-dominant forearm)
* Self-reported use of opioids in last week
* Comorbid condition for which exercise is deemed unsafe by a physician or the (Physical Activity Readiness Questionnaire+) PARQ+
* unable to safely ambulate on a treadmill

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Thresholds (PPT) | Before and after the intervention at baseline
  A pressure algometer is applied 3 times to 2 sites: the dominant quadriceps and deltoid using the Force Ten FDX pressure gauge (Wagner Instruments, Greenwich, CT). The pressure at which the participant reports pain is recorded and averaged over the three trials. Higher PPTs represent less pain sensitivity.
Offset Analgesia Response | Before and after the intervention at baseline
  Percent decrease in pain reported between T2 and T3 interval of the offset analgesia test. Higher values represent greater pain inhibition.
Temporal Summation of Heat Pain | Before and after the intervention at baseline
  To evaluate constant noxious heat pain summation, a noxious heat stimulus (60/100 on a visual analogue scale) is held for 60 seconds. Temporal summation is defined by an exponential increase in pain at the test end relative to the start; greater values represent greater pain facilitation.

SECONDARY OUTCOMES:
Fitkids Treadmill Test | Single measurement at baseline
  Time to exhaustion (TTE) on the FTT provides an objective, norm-referenced marker of aerobic capacity in youth and is defined as the total time completed on the test, excluding the warm-up and cool-down phases. Data recorded includes TTE, rate of perceived exertion (Borg Scale), and maximum heart rate. Successful completion of the exercise session will be defined as achievement of > 85% age-predicted maximum heart rate. Greater TTE represents greater aerobic fitness.
Functional Disability Inventory | Single measurement at baseline
  15-item Likert scale of pain related disability. Higher scores represent greater disability.
Tampa Kinesiophobia Scale | Single measurement at baseline
  Likert type scale of movement related fear. Higher scores indicate greater fear.
Pain Catastrophizing Scale | Single assessment at baseline
  Likert type patient reported outcome of worry related to pain. HIgher score represent greater worries related to pain.
Fear of Pain Questionnaire Child | Single assessment at baseline.
  Patient reported outcome of pain related fear. Higher scores reflect greater fear.
PROMIS Pediatric Pain Interference - Short Form 8a | Single assessment at baseline
  Patient reported outcome of pain impact on life. Higher score reflect greater pain interference.
Central Sensitization Inventory | Single assessment at baseline.
  Patient reported outcome of the frequency of symptoms commonly experienced by persons with chronic pain. Higher score represent greater central sensitization.
Numeric Pain Rating Scale | Baseline - before and after intervention
  Self-reported pain intensity on an 11-point likert scale. Higher scores represent greater pain intensity.
Highly Sensitive Child Scale | Single measurement at baseline
  Patient reported outcome of sensitivity to common daily sensory stimuli. Higher scores represent greater sensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital at 2 Brookline Place, Brookline, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD not covered by the informed consent process will not be shared for privacy reasons.

REFERENCES:
- [Background] Chambers CT, Dol J, Tutelman PR, Langley CL, Parker JA, Cormier BT, Macfarlane GJ, Jones GT, Chapman D, Proudfoot N, Grant A, Marianayagam J. The prevalence of chronic pain in children and adolescents: a systematic review update and meta-analysis. Pain. 2024 Oct 1;165(10):2215-2234. doi: 10.1097/j.pain.0000000000003267. Epub 2024 May 15. PMID 38743558
- [Background] Shulman J, Zurakowski D, Keysor J, Jervis K, Sethna NF. Offset analgesia identifies impaired endogenous pain modulation in pediatric chronic pain disorders. Pain. 2020 Dec;161(12):2852-2859. doi: 10.1097/j.pain.0000000000001984. PMID 32658151
- [Background] Rice D, Nijs J, Kosek E, Wideman T, Hasenbring MI, Koltyn K, Graven-Nielsen T, Polli A. Exercise-Induced Hypoalgesia in Pain-Free and Chronic Pain Populations: State of the Art and Future Directions. J Pain. 2019 Nov;20(11):1249-1266. doi: 10.1016/j.jpain.2019.03.005. Epub 2019 Mar 21. PMID 30904519
- [Background] Grill JD, Coghill RC. Transient analgesia evoked by noxious stimulus offset. J Neurophysiol. 2002 Apr;87(4):2205-8. doi: 10.1152/jn.00730.2001. PMID 11929939
- [Background] Stolzman S, Danduran M, Hunter SK, Bement MH. Pain Response after Maximal Aerobic Exercise in Adolescents across Weight Status. Med Sci Sports Exerc. 2015 Nov;47(11):2431-40. doi: 10.1249/MSS.0000000000000678. PMID 25856681
- [Background] Stolzman S, Bement MH. Does Exercise Decrease Pain via Conditioned Pain Modulation in Adolescents? Pediatr Phys Ther. 2016 winter;28(4):470-3. doi: 10.1097/PEP.0000000000000312. PMID 27661245